CLINICAL TRIAL: NCT04703244
Title: Development of Patient Derived Xenografts (PDX) in Patients With Breast Cancer Who Have Residual Disease After Neoadjuvant Systemic Therapy
Brief Title: Development of Patient Derived Xenografts (PDX) in Patients With Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1933
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Residual
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: chemotherapy or endocrine therapy for breast cancer — Collect blood and leftover surgical tissue from patients with breast cancer remaining after chemotherapy or endocrine therapy is completed.

SUMMARY:
Breast cancer patients who undergo neoadjuvant systemic therapy and have residual breast cancer identified at the time of surgery exhibit a high (>50%) risk of future life-threatening recurrences and death.

DETAILED DESCRIPTION:
This study is being done to collect blood and leftover surgical tissue from patients with breast cancer remaining after chemotherapy or endocrine therapy is completed. We will use the blood and tissue for future studies. These studies will try to find ways to treat future breast cancer patients.

Because there is cancer left in your body after breast cancer treatment is finished, we think the cancer may be different than other cancers. Tissue from surgery will be used to try to grow that kind of cancer in the lab so we can find out more about it and how to treat it.

Blood samples will be used to look at measurements of biomarkers to see how this cancer is different and seek new ways to identify and treat it.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of invasive breast cancer treated with neoadjuvant systemic therapy.
* Surgically resectable disease following neoadjuvant systemic treatment.
* At least one of the following must be true:

  1. Received at least 2 weeks of neoadjuvant endocrine therapy
  2. Received at least 2 months of neoadjuvant chemotherapy with suggestion of residual disease on imaging
  3. Began neoadjuvant chemotherapy or endocrine therapy but discontinued due to evidence of progressive disease by MRI, ultrasound, or physical examination
* Provide written informed consent.
* Willing to return to enrolling institution for breast cancer surgery.
* Willingness to provide mandatory blood specimens for future research on breast cancer at Mayo Clinic.
* Willingness to provide mandatory tissue specimens for future research on breast cancer at Mayo Clinic.
* Willingness to provide mandatory tissue specimens for the generation of PDX and organoids to be used future research on breast cancer at Mayo Clinic.

Exclusion Criteria:

* Ineligible for surgery.
* History of prior malignancy <3 years prior to registration. Exceptions for non-melanoma skin cancer, papillary thyroid cancer, non-invasive cancer (e.g., carcinoma in situ of the cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have completed neoadjuvant systemic therapy who have residual disease on post-neoadjuvant imaging and are planning surgical resection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2041-01-15 (Estimated); Study Completion 2042-01-15 (Estimated)

PRIMARY OUTCOMES:
Generate patient derived xenografts (PDX) and organoids from breast cancer patients with residual disease after neoadjuvant therapy | Up to 12 months until death or a maximum of 20 years post registration

SECONDARY OUTCOMES:
Utilize patient derived xenografts (PDX) models to study new drugs/drug combinations | Up to 12 months until death or a maximum of 20 years post registration
Utilize patient derived xenografts (PDX) models to identify mechanisms of treatment resistance | Up to 12 months until death or a maximum of 20 years post registration
Correlate the association between Cell Free DNA (cfDNA), Circulating Tumor Cells (CTCs) and circulating immune cell subpopulations (as measured by CyTOF) with residual cancer burden | Up to 12 months until death or a maximum of 20 years post registration
Correlate the association between Cell Free DNA (cfDNA) with residual cancer burden | Up to 12 months until death or a maximum of 20 years post registration
Correlate the association between Circulating Tumor Cells (CTCs) with residual cancer burden | Up to 12 months until death or a maximum of 20 years post registration
Correlate the association between circulating immune cell subpopulations (as measured by Cytometry by time-of-flight (CyTOF) with residual cancer burden | Up to 12 months until death or a maximum of 20 years post registration
Generate autologous co-culture systems of peripheral blood immune cells and breast cancer tumor cells to study the endogenous antitumor immune response | Up to 12 months until death or a maximum of 20 years post registration

CONTACTS AND LOCATIONS:
Overall Officials: Judy C. Boughey, M.D., Principal Investigator — Mayo Clinic; Matthew P. Goetz, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No